CLINICAL TRIAL: NCT03943511
Title: A Randomized Study Evaluating Patients Discharged With Indwelling Chest Tube and Valve
Brief Title: Discharged With Indwelling Chest Tube and Valve
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low accrual, end of funding
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, K Robert Shen, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 17-007774
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Prolonged Air Leak
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Active Comparator): Oral Antibiotics
  Interventions: Other: Oral Antibiotics-Close Monitoring
- Group 2 (Active Comparator): Standard of Care
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Oral Antibiotics-Close Monitoring — To receive oral antibiotics and close monitoring, defined as twice weekly telephone calls by a member of the care team, of their chest tube and valve.
  Arms: Group 1
Other: Standard of Care — No calls from the care team but waiting for the subject to contact the care team when the air leak has stopped.
  Arms: Group 2

SUMMARY:
This study is a multicenter, randomized trial for the treatment of subjects discharging from the hospital with a chest tube and valve in place. Subjects will be randomized to receive oral antibiotics and close monitoring, defined as twice weekly telephone calls by a member of the care team, of their chest tube and valve or standard of care, defined as no calls from the care team but waiting for the subject to contact the care team when the air leak has stopped.

DETAILED DESCRIPTION:
This study is a multicenter, randomized trial for the treatment of subjects discharging from the hospital with a chest tube and valve in place. Subjects will be screened prior to discharging from the hospital and interested qualified subjects will be consented and offered participation in this trial. Once consent has been obtained the subject will be randomized to receive oral antibiotics and close monitoring, defined as twice weekly telephone calls by a member of the care team, of their chest tube and valve or standard of care, defined as no calls from the care team but waiting for the subject to contact the care team when the air leak has stopped. The subject will be followed until they have their chest tube removed.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Male and Female
* Consultation with a thoracic surgeon
* Discharge from the hospital with a chest tube and valve in place
* Subject is able to understand the study procedures and provide informed consent.

Exclusion Criteria:

* Pregnancy
* Allergy to Keflex and Clindamycin
* Special consideration should be taken in enrolling subjects with preexisting conditions that can be exacerbated by antibiotic use but are allowed at the discretion of the treating physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-07 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Change in empyema in patient's discharging with an indwelling chest tube and valve. | 30 days post discharge
  The proportion of patients having 30-day empyema in the two treatment arms will be estimated and reported.

SECONDARY OUTCOMES:
Change of 30-day readmission in patient's discharging with an indwelling chest tube and valve. | 30 days post discharge
  The proportion of patients having a 30-day readmission in the two treatment arms will be estimated and reported.

CONTACTS AND LOCATIONS:
Overall Officials: K. Robert Shen, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Rush University Medical Center, Chicago, Illinois
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials